CLINICAL TRIAL: NCT05694091
Title: Correlation of Perioperative Brain Metabolites With Postoperative Delirium in Elderly Oral Craniomaxillofacial Surgery Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Other Study IDs: SH9H-2022-T331-1
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2022-11

CONDITIONS: Delirium in Old Age
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Blood Specimen Collection; Urination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients in the control group were followed up without delirium postoperatively.: If the 3D-CAM scale all show a negative resluts
  Interventions: Other: Collecting clinical data, blood gas data, Magnetic Resonance Spectroscopy (MRS) data and blood,urine, and feces sample
- Patients in the case group were followed up with delirium postoperatively.: If the 3D-CAM assessment is positive at any time point after surgery
  Interventions: Other: Collecting clinical data, blood gas data, Magnetic Resonance Spectroscopy (MRS) data and blood,urine, and feces sample

INTERVENTIONS:
Other: Collecting clinical data, blood gas data, Magnetic Resonance Spectroscopy (MRS) data and blood,urine, and feces sample — Collecting clinical data(before induction of anesthesia and first day after surgery), blood gas data(before induction of anesthesia and first day after surgery) ，MRS data (not more than 24h after surgery）and blood,urine, and feces sample （before induction of anesthesia and first day, third day and 7th day after surgery）

SUMMARY:
In view of the increasingly severe aging situation in China, the perioperative brain health of elderly patients has received increasing attention. Postoperative delirium (POD) is a common postoperative complication characterized by acute consciousness and cognitive dysfunction. The incidence of POD in elderly patients undergoing elective non cardiac surgery is 20%~45%, which often indicates poor cognitive recovery and becomes a heavy burden for family and society. Although the weight of human brain only accounts for 2% of body weight, the oxygen consumption accounts for 20% of the total oxygen consumption of the whole body. On July 2, 2022, the British Journal of Anaesthesia (Chinese Academy of Sciences Division 1, Anesthesiology Division 1, IF11.719), the top international Journal in the field of anesthesiology, published the scientific research achievements of the first author of the applicant. It was found for the first time that sevoflurane, the most commonly used inhalation anesthetic in clinical practice, can cause the activation of glycolysis and the increase of lactic acid in the brain of elderly non-human primate marmosets, which suggests that general anesthetics will affect brain metabolism in the perioperative period. Therefore, we hypothesized that perioperative changes in brain metabolism might be related to the occurrence of POD in elderly patients. The purpose of this study was to study the relationship between the changes of brain metabolites and POD during perioperative period by noninvasive monitoring of the characteristics of brain tissue metabolites 24 hours before and 24 hours after the operation with hydrogen ion proton magnetic resonance spectroscopy (1-HMRS). In order to complete this purpose, this study plans to collect subjects aged 65~90 years who are scheduled to undergo oral and maxillofacial surgery under general anesthesia. The changes of brain metabolites before and after operation were collected by 1-HMRS, and the postoperative delirium related scale was evaluated to analyze the relationship between perioperative changes of brain metabolites and POD.

ELIGIBILITY:
Inclusion Criteria:

* The ASA grade of the subject is Ⅰ - Ⅲ;
* 65-90 years old;
* Oral craniomaxillofacial surgery under combined general anesthesia

Exclusion Criteria:

* The following medical devices have been installed in the body or are to be installed or implanted in the hospital: various cardiac pacemakers; Metal implants (non titanium), ferromagnetic vascular clips in the body
* The patient is left-handed;
* Patients with claustrophobia;
* People with vision and hearing impairment, illiterate or difficult to communicate;
* The operation plan includes patients with tracheotomy or postoperative catheterization;
* Refusing to sign the clinical trial consent form.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Our research is a single center, nested case-control study. Preoperatively collect the information of the elderly patients 65-90 years old without undergoing craniocerebral operations, including the vital signs, the examination reports and other related data after excluding the factors that can't be included in the group. The patients' health scales and delirium scales were evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
3D-CAM (3-minute Diagnostic Interview for Confusion Assessment Method) scale | 1 day after surgery
  3D-CAM higher means worse
3D-CAM (3-minute Diagnostic Interview for Confusion Assessment Method) scale | 2 day after surgery
  3D-CAM higher means worse
3D-CAM (3-minute Diagnostic Interview for Confusion Assessment Method) scale | 3 day after surgery
  3D-CAM higher means worse
3D-CAM (3-minute Diagnostic Interview for Confusion Assessment Method) scale | 4 day after surgery
  3D-CAM higher means worse
3D-CAM (3-minute Diagnostic Interview for Confusion Assessment Method) scale | 5 day after surgery
  3D-CAM higher means worse
3D-CAM (3-minute Diagnostic Interview for Confusion Assessment Method) scale | 6 day after surgery
  3D-CAM higher means worse
3D-CAM (3-minute Diagnostic Interview for Confusion Assessment Method) scale | 7 day after surgery
  3D-CAM higher means worse

SECONDARY OUTCOMES:
MOCA(Montreal Cognitive Assessment) scale | 1 day after surgery
  MOCA higher means better
MOCA(Montreal Cognitive Assessment) scale | 3 day after surgery
  MOCA higher means better
MOCA(Montreal Cognitive Assessment) scale | 7 day after surgery
  MOCA higher means better
MMSE (mini-mental state examiniation) scale | 1 day after surgery
  MMSE higher means better
MMSE (mini-mental state examiniation) scale | 3 day after surgery
  MMSE higher means better
MMSE (mini-mental state examiniation) scale | 7 day after surgery
  MMSE higher means better

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jiang, Doctor, Study Director — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai 9Th Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No